CLINICAL TRIAL: NCT04358471
Title: A Phase 2 Multi-Center Trial Evaluating Intravitreal AAVCAGsCD59 Compared to Sham Injection for the Treatment of Advanced Dry Age-Related Macular Degeneration (AMD) With Geographic Atrophy (GA)
Brief Title: Intravitreal AAVCAGsCD59 for Advanced Dry Age-related Macular Degeneration (AMD) With Geographic Atrophy (GA)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The AAVCAGsCD59 asset has been transferred to Janssen Research and Development LLC
Sponsor: Hemera Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMR-2001
Record Dates: First submitted 2020-03-22; First posted 2020-04-24 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Dry Age-related Macular Degeneration; Geographic Atrophy; Gene Therapy; Intravitreal Injection
MeSH Terms: conditions — Geographic Atrophy | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to low dose AAVCAGsCD59, high dose AAVCAGsCD59, or sham arm.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Intravitreal AAVCAGsCD59 1.071x10e12 vg Injection (Active Comparator): Intravitreal AAVACGsCD59 at a dose of 1.071x10e12 vg administered once on Day 0
  Interventions: Biological: Intravitreal AAVCAGsCD59
- Intravitreal AAVCAGsCD59 3.56x10e11 vg Injection (Active Comparator): Intravitreal AAVACGsCD59 at a dose of 3.56x10e11 vg administered once on Day 0
  Interventions: Biological: Intravitreal AAVCAGsCD59
- Sham Intravitreal Injection (Sham Comparator): Intravitreal Sham injection administered once on Day 0
  Interventions: Other: Intravitreal Sham Injection

INTERVENTIONS:
Biological: Intravitreal AAVCAGsCD59 — AAVCAGsCD59 is administered as an intravitreal injection in the enrolled eye
  Other Names: HMR59
  Arms: Intravitreal AAVCAGsCD59 1.071x10e12 vg Injection; Intravitreal AAVCAGsCD59 3.56x10e11 vg Injection
Other: Intravitreal Sham Injection — Sham injection mimics a real injection in the enrolled eye
  Other Names: Sham
  Arms: Sham Intravitreal Injection

SUMMARY:
Patients with advanced dry AMD with GA meeting inclusion criteria will be randomized in one eye in a 1:1:1 ratio comparing intravitreal high or low dose AAVCAGsCD59 with a sham injection. All enrolled subjects will be followed for 24 months to evaluate reduction in GA growth and safety of intravitreal AAVCAGsCD59.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced dry AMD with GA in the study eye
2. BCVA in the study eye of 80 or less ETDRS letters (Snellen equivalent 20/25 or worse)
3. Total cumulative GA lesion size 2.5 mm2 to 12.5 mm2 in the study eye as confirmed by the reading center during the Screening Period.

Exclusion Criteria:

1. GA secondary to non-AMD etiologies in the study eye (i.e. myopia, inherited retinal diseases).
2. GA associated with the presence of an RPE rip.
3. GA contiguous with peripapillary atrophy.
4. Active CNV secondary to wet AMD in the study eye and currently receiving anti-VEGF ocular treatment within the previous 18 months.
5. Subretinal fibrosis in the macula from CNV both clinically and imaged on SD-OCT in the macula.
6. Previous macular laser photocoagulation (i.e. focal or grid laser for macular edema), photodynamic therapy (PDT), ocular/orbital radiation, laser to CNV, or subretinal surgery for CNV in the study eye.
7. History of conditions in the study eye which might alter visual acuity or interfere with study testing including proliferative diabetic retinopathy (PDR), clinically significant macular edema (CSME), central retinal vein occlusion (CRVO), hemi retinal vein occlusion (HRVO), macular branch retinal vein occlusion, and optic neuropathy.
8. Active uncontrolled glaucoma with at least one of the following: IOP>30 mmHg despite maximum medical treatment with glaucoma medications, cup-to-disc ratio of >0.9, visual field defects secondary to glaucoma that involve the macula, or optic atrophy from glaucoma.
9. Active acute or chronic infectious uveitis, retinitis, or conjunctivitis (excluding blepharitis)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-31 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the change in Geographic Atrophy area (mm2) measured at Day 0 and compared to the measurement at Month 24 | 24 Months
  Geographic atrophy will be measured based on imaging of the retina

SECONDARY OUTCOMES:
Incidence of conversion from dry to wet age-related macular degeneration | 24 Months
  Measure the number of treated eyes in the sham and AAVCAGsCD59-treated arms that convert from dry to wet age-related macular degeneration
Change in visual acuity of the AAVCAGsCD59 treated eye | 24 Months
  Visual acuity measured on an Early Treatment Diabetic Retinopathy Study (ETDRS) chart will be compared at Day 0 and Month 24

IPD SHARING:
Plan to Share IPD: No